CLINICAL TRIAL: NCT04562792
Title: A Pilot Study of Targeted Daunorubicin Dosing to Overcome Chemotherapeutic Resistance in Children With Relapsed or Refractory Acute Leukemia
Brief Title: Low Dose Daunorubicin in Pediatric Relapsed/Refractory Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001114
Record Dates: First submitted 2020-08-28; First posted 2020-09-24 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Relapsed Pediatric ALL; Relapsed Pediatric AML; Refractory Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with relapsed/refractory ALL and AML (Experimental): Patients in this arm will receive daunorubicin 6.75mg/m2 daily for 5 consecutive days.
  Interventions: Drug: Daunorubicin

INTERVENTIONS:
Drug: Daunorubicin — Eligible patients with relapsed and/or refractory acute leukemia will receive daunorubicin 6.75mg/m2 daily for 5 consecutive days.

SUMMARY:
In this pilot study, eligible pediatric patients will be treated with 5 consecutive days of low dose daunorubicin. All patients who receive low dose daunorubicin will be evaluated daily for potential toxicity during those 5 days. Once the patient has received 5 doses of daunorubicin, subsequent therapy will be at the discretion of the primary oncology team.

DETAILED DESCRIPTION:
Cancer remains the number one cause of non-accidental death in children with leukemia being the most common type of childhood cancer. Although cure rates for pediatric leukemia have greatly improved over the last few years, relapsed disease still carries a poor prognosis. Outcomes for children with multiply relapsed leukemia are dismal ranging from a remission rate of 25% in AML after 2 relapses falling to 17% after 3 or more relapses and 44% in ALL after 2 relapses and 27% after 3 or more relapses.

Leukemia stem cells that are resistant to chemotherapy primarily contribute to treatment failure and targeting these cells remains a challenge. Anthracyclines such as daunorubicin and doxorubicin have been the mainstays of childhood leukemia therapy for over 50 years. Prior investigations found that very low doses, significantly less than traditionally given, of doxorubicin and daunorubicin inhibit the interaction of Akt and beta catenin pathways which is known to drive the development of leukemia stem cells and chemoresistance. Mice models showed that treatment with these very low dose anthracyclines does not suppress the immune system but rather expands cancer targeting T cells while inhibiting populations known to help cancer cells evade the immune system. In addition, targeted treatment reduced immune checkpoint expression, a known cause of resistance, on leukemia stem cells, thus further sensitizing them to cytotoxic T cells. Standard doses of anthracyclines suppress hematopoiesis and in turn the immune system and thus do not permit the expression of these immunologic benefits.

Patients with relapsed and/or refractory acute lymphoblastic leukemia or acute myeloid leukemia, ages 1-21 years, will be approached to participate in this study. These patients must have pathologically confirmed ALL or AML, whose disease is refractory to two induction therapeutic attempts, or who are in 2nd or greater relapse, or who are in 1st relapse or refractory to a single therapeutic attempt but are unable to receive intensive therapy due to other comorbidities. Patients will receive daunorubicin at 6.75mg/m2 daily for 5 consecutive days for a total dose of 33.75mg/m2.

The primary objective of this study is to assess the feasibility and tolerability of low dose daunorubicin. Another objective of the study is to validate if T cell based immune responses against chemoresistant leukemia stem cells are stimulated at these lower doses of daunorubicin, in hopes to provide preliminary pediatric data for further research with the hypothesis being that targeted anthracycline treatment does in fact stimulate T cell based immune responses against chemoresistant leukemia stem cells. Samples will be analyzed by flow cytometry for stem cell and immune markers. The third primary objective is to identify pro vs anti-cancer cellular immune responses of targeted anthracycline treatment in these patients. The mechanism of low dose DNR treatment on activating immunogenic cell death (ICD) will be investigated by determining relative levels of damage-associated molecular patterns. The tumorigenic capacity of resistant populations such as LSCs expressing high levels of immune checkpoints will be tested. The secondary objective of this study is to evaluate the pharmacokinetic parameters of low dose daunorubicin in children with relapsed/refractory AML and ALL. Blood samples for evaluation of low dose daunorubicin pharmacokinetics (area under the time concentration curve, maximum concentration, elimination half-life, clearance) will be drawn prior to dosing and 5min, 20min, 40min, 1hr, 2hrs, 4hrs, 8hrs, and 24hrs only after the first day of dosing.

Once the patient has received 5 doses of daunorubicin, subsequent therapy will be at the discretion of the primary oncology team.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed ALL or AML, whose disease is refractory to two induction therapeutic attempts, or who are in 2nd or greater relapse, or who are in 1st relapse or refractory to a single therapeutic attempt but are unable to receive intensive therapy at the time of consent.
* All prior upfront therapies including bone marrow transplant are acceptable. Pulse steroids (of 5 days duration or less in the prior month) administered as part of a routine maintenance therapy are acceptable.
* Age 1 to 21 years of age, inclusive
* Established central catheter IV access

Exclusion Criteria:

* Females who are known to be pregnant or lactating
* Any Grade 3 or higher Cardiac Disorder per CTCAE version 5
* Patients with echocardiographic evidence of cardiomyopathy (shortening fraction <27% or ejection fraction <50%)
* Uncontrolled sepsis
* Absolute Blast Count >50 x10(3)/mcL at enrollment or on day 1 of study
* Direct hyperbilirubinemia >5mg/dL
* Grade 3 or higher anaphylaxis to daunorubicin
* Non-English speaking
* Patients, who in the opinion of the PI, are unable to tolerate any study-specific procedures
* Patients who have received cyclosporine, tacrolimus or other agents to prevent or treat graft-vs-host disease post bone marrow transplant in the last 14 days
* Concurrent investigational drugs or other chemotherapeutic agents (excluding hydroxyurea), immunotherapies or biosimilars during the 5 days of daunorubicin.
* Prior cumulative doses of anthracyclines will not be an exclusion regardless of the total cumulative dose previously received.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandni Dargan, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward E, DeSantis C, Robbins A, Kohler B, Jemal A. Childhood and adolescent cancer statistics, 2014. CA Cancer J Clin. 2014 Mar-Apr;64(2):83-103. doi: 10.3322/caac.21219. Epub 2014 Jan 31. PMID 24488779
- [Background] Nguyen K, Devidas M, Cheng SC, La M, Raetz EA, Carroll WL, Winick NJ, Hunger SP, Gaynon PS, Loh ML; Children's Oncology Group. Factors influencing survival after relapse from acute lymphoblastic leukemia: a Children's Oncology Group study. Leukemia. 2008 Dec;22(12):2142-50. doi: 10.1038/leu.2008.251. Epub 2008 Sep 25. PMID 18818707
- [Background] Borowitz MJ, Devidas M, Hunger SP, Bowman WP, Carroll AJ, Carroll WL, Linda S, Martin PL, Pullen DJ, Viswanatha D, Willman CL, Winick N, Camitta BM; Children's Oncology Group. Clinical significance of minimal residual disease in childhood acute lymphoblastic leukemia and its relationship to other prognostic factors: a Children's Oncology Group study. Blood. 2008 Jun 15;111(12):5477-85. doi: 10.1182/blood-2008-01-132837. Epub 2008 Apr 3. PMID 18388178
- [Background] Armenian SH. Improving screening practices in childhood cancer survivors at risk for treatment-related heart failure. J Clin Oncol. 2014 Dec 10;32(35):3923-5. doi: 10.1200/JCO.2014.58.5562. Epub 2014 Nov 3. No abstract available. PMID 25366690
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Kawashima T, Hudson MM, Meadows AT, Friedman DL, Marina N, Hobbie W, Kadan-Lottick NS, Schwartz CL, Leisenring W, Robison LL; Childhood Cancer Survivor Study. Chronic health conditions in adult survivors of childhood cancer. N Engl J Med. 2006 Oct 12;355(15):1572-82. doi: 10.1056/NEJMsa060185. PMID 17035650
- [Background] Reulen RC, Winter DL, Frobisher C, Lancashire ER, Stiller CA, Jenney ME, Skinner R, Stevens MC, Hawkins MM; British Childhood Cancer Survivor Study Steering Group. Long-term cause-specific mortality among survivors of childhood cancer. JAMA. 2010 Jul 14;304(2):172-9. doi: 10.1001/jama.2010.923. PMID 20628130
- [Background] Blanco JG, Sun CL, Landier W, Chen L, Esparza-Duran D, Leisenring W, Mays A, Friedman DL, Ginsberg JP, Hudson MM, Neglia JP, Oeffinger KC, Ritchey AK, Villaluna D, Relling MV, Bhatia S. Anthracycline-related cardiomyopathy after childhood cancer: role of polymorphisms in carbonyl reductase genes--a report from the Children's Oncology Group. J Clin Oncol. 2012 May 1;30(13):1415-21. doi: 10.1200/JCO.2011.34.8987. Epub 2011 Nov 28. PMID 22124095
- [Background] van Nimwegen FA, Ntentas G, Darby SC, Schaapveld M, Hauptmann M, Lugtenburg PJ, Janus CPM, Daniels L, van Leeuwen FE, Cutter DJ, Aleman BMP. Risk of heart failure in survivors of Hodgkin lymphoma: effects of cardiac exposure to radiation and anthracyclines. Blood. 2017 Apr 20;129(16):2257-2265. doi: 10.1182/blood-2016-09-740332. Epub 2017 Jan 31. PMID 28143884
- [Background] Felker GM, Thompson RE, Hare JM, Hruban RH, Clemetson DE, Howard DL, Baughman KL, Kasper EK. Underlying causes and long-term survival in patients with initially unexplained cardiomyopathy. N Engl J Med. 2000 Apr 13;342(15):1077-84. doi: 10.1056/NEJM200004133421502. PMID 10760308
- [Background] Huang J, Nguyen-McCarty M, Hexner EO, Danet-Desnoyers G, Klein PS. Maintenance of hematopoietic stem cells through regulation of Wnt and mTOR pathways. Nat Med. 2012 Dec;18(12):1778-85. doi: 10.1038/nm.2984. Epub 2012 Nov 11. PMID 23142822
- [Background] Korkaya H, Paulson A, Charafe-Jauffret E, Ginestier C, Brown M, Dutcher J, Clouthier SG, Wicha MS. Regulation of mammary stem/progenitor cells by PTEN/Akt/beta-catenin signaling. PLoS Biol. 2009 Jun 2;7(6):e1000121. doi: 10.1371/journal.pbio.1000121. Epub 2009 Jun 2. PMID 19492080

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Low Dose Daunorubicin Feasbility as Assessed by Absolute Blast Count
Description: Feasibility failure due to progressive leukemia is defined as a rise in absolute blast count (ABC) of >10,000/day on two consecutive days that continues to increase >10,000/day after starting hydroxyurea.
Time Frame: 24 months
Population: Data collected but analysis not performed due to small number of participants and inability to run analysis without more samples
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 1
Participants
  Patients with a rise in absolute blast count (ABC) of >10,000/day on two consecutive days | 0
  Patients without a rise in absolute blast count (ABC) of >10,000/day on two consecutive days | 1

2. Primary Outcome: Incidence of Low Dose Daunorubicin Feasbility as Assessed by Extramedullary Leukemia Progression
Description: Low dose daunorubicin will also be deemed not feasible if there is evidence of progression of extramedullary leukemia such progression of chloroma or leukemia cutis. or if the patient experiences uncontrollable nausea and/or vomiting.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 1
Participants
  Patients with evidence of progression of extramedullary leukemia | 0
  Patients without evidence of progression of extramedullary leukemia | 1

3. Primary Outcome: Incidence of Low Dose Daunorubicin Feasbility as Assessed by Patient Symptoms
Description: Low dose daunorubicin will also be deemed not feasible if the patient experiences uncontrollable nausea and/or vomiting.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 1
Participants
  Uncontrollable Nausea or Vomiting | 0
  Patients with no uncontrollable nausea or vomiting | 1

4. Primary Outcome: T-cell Based Immune Responses Against Chemoresistant Leukemia Stem Cells (LSC) Are Stimulated at Lower Doses of Daunorubicin to Provide Preliminary Data for Further Research.
Description: Leukemia stem cells (LSCs) are known to be resistant to chemotherapy which may lead to treatment failure. In vitro studies have shown that targeted anthracycline treatment reduces immune checkpoint expression on LSCs, potentially sensitizing LSCs to cytotoxic T-cells. This will be measured in our study.
Time Frame: 24 months
Population: This particular outcome measure requires analysis to be run in the laboratory. This was not performed and therefore there is not data to report.
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 0

5. Primary Outcome: The Pro- vs. Anti-cancer Cellular Immune Response of Targeted Anthracycline Treatment in Patients With Relapsed/Refractory Acute Leukemia
Description: Chemotherapy is typically administered at maximum tolerated doses which leads to secondary immunosuppression. In other words, beneficial immunologic side effects can be weakened if chemotherapy is given at high doses. The Wnt pathway (which plays a key role in chemoresistance of LSCs) reduces T cell recruitment to tumors. Available data in murine models indicates that targeted anthracycline treatment expands cancer-targeting T-cells while inhibiting populations known to help cancer cells evade the immune system. This will be measured in our study.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 0

6. Secondary Outcome: Pharmacokinetic Parameters of Low Dose Daunorubicin in Children With Relapsed/Refractory AML and ALL as Assessed by Maximum Concentration.
Description: Serial daunorubicin levels for evaluation of maximum concentration will be drawn prior to infusion and at 5, 20 and 40 minutes and at hours 1,2,4,8 and 24 post infusion.
Time Frame: 24 months
Population: One patient analyzed.
Measure: Number; unit: ng/mL
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 1
ng/mL | 18.7

7. Secondary Outcome: Pharmacokinetic Parameters of Low Dose Daunorubicin in Children With Relapsed/Refractory AML and ALL as Assessed by Time at Maximum Concentration.
Description: Serial daunorubicin levels for evaluation of time at maximum concentration will be drawn prior to infusion and at 5, 20 and 40 minutes and hours 1,2,4,8 and 24 post infusion.
Time Frame: 24 months
Population: One patient analyzed.
Measure: Number; unit: hour
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 1
hour | 0.33333

8. Secondary Outcome: Pharmacokinetic Parameters of Low Dose Daunorubicin in Children With Relapsed/Refractory AML and ALL as Assessed by Area Under the Curve.
Description: Serial daunorubicin levels for evaluation of exposure by measuring area under the curve will be drawn prior to infusion and at 5, 20 and 40 minutes and hours 1,2,4,8 and 24 post infusion.
Time Frame: 24 months
Population: One patient analyzed.
Measure: Number; unit: hr*ng/mL
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 1
hr*ng/mL | 20.889865

9. Secondary Outcome: Pharmacokinetic Parameters of Low Dose Daunorubicin in Children With Relapsed/Refractory AML and ALL as Assessed by Elimination Half-life
Description: Serial daunorubicin levels for evaluation of exposure by measuring elimination half-life will be drawn prior to infusion and at 5, 20 and 40 minutes and hours 1,2,4,8 and 24 post infusion.
Time Frame: 24 months
Population: One patient analyzed.
Measure: Number; unit: hour
Arm/Group | Patients With Relapsed/Refractory ALL and AML
Number analyzed (Participants) | 1
hour | 1.8588

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Patients With Relapsed/Refractory ALL and AML
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT04562792/Prot_001.pdf